CLINICAL TRIAL: NCT06027736
Title: The Effectiveness of Pharmacist-led Educational Model in Patients With Allergic Rhinitis in a Malaysian Tertiary Hospital: A Randomised Control Trial Protocol (AR-PRISE RCT)
Brief Title: The Effectiveness of Pharmacist-led Educational Model in Patients With Allergic Rhinitis
Acronym: AR-PRISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Chee Ping Chong (Other)
Collaborators: Hospital Raja Permaisuri Bainun (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Chee Ping Chong, Senior Lecturer, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NMRR ID-22-01621-I1W (IIR)
Record Dates: First submitted 2023-08-23; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Allergic Rhinitis; Pharmaceutical Care; Pharmaceutical Services
Keywords: Allergic rhinitis; Pharmacist; Education; Pharmaceutical services
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: pharmacist-led education
- Control group (No Intervention)

INTERVENTIONS:
Other: pharmacist-led education — A patient education protocol and an algorithm of pharmaceutical care in managing allergic rhinitis.
  Arms: Intervention group

SUMMARY:
Allergic rhinitis is a chronic respiratory disorder affecting patients' quality of life and work performance. Pharmacists are identified as suitable professionals to deliver patient education and pharmaceutical care in managing allergic rhinitis (AR) patients. Local clinical practice guidelines in Malaysia are lacking, especially in pharmaceutical care in public healthcare institutions. This study protocol describes a randomised control trial (RCT) that aims to determine the effectiveness of a pharmacist-led educational model in managing AR (AR-PRISE Model) compared to standard pharmaceutical care. The AR-PRISE model delivers patient educational material (video) and an algorithm for pharmaceutical care.

DETAILED DESCRIPTION:
This is a six-month, single-centre, prospective, randomised, two-arm, and parallel-group controlled trial. This trial recruits patients attending a tertiary hospital's otorhinolaryngology outpatient clinics. The participants are randomised into the control or intervention groups at 1:1 using permuted block randomisation. Each group required 77 participants. The control group will receive standard pharmaceutical care. The intervention group will receive pharmacist-led education according to the AR-PRISE model. Both groups will be assessed for the middle turbinate endoscopy findings, disease severity, knowledge level, symptom control, medication adherence, and quality of life (QoL) at baseline and end-of-study follow-up (Day 180±7). Depending on the feasibility at Day 60±7 and 120±7, they will be followed up virtually or face-to-face. During the intermediate follow-up, the participants will be assessed for symptom control, medication adherence, and QoL. The intention-to-treat analysis will include all participants assigned to each group. An Independent T-Test compares the mean difference in knowledge level between the two groups. A two-way repeated measure ANOVA analysis will be employed to determine between-group differences for scores of symptom control, adherence rate, and QoL. A one-way repeated measure ANOVA will be performed for within-group analysis. A P-value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients include an aged 18 to 80, Malaysian, diagnosed with allergic rhinitis, and capable of reading and writing in English or Malay, who attend the otorhinolaryngology outpatient clinic at Raja Permaisuri Bainun Hospital.

Exclusion Criteria:

* Patients who are pregnant, lactating, or have a comorbid diagnosis of chronic rhinosinusitis will be excluded.
* Patients having psychiatric problems, dementia, terminal illnesses, comorbidities, post-COVID-19 conditions with symptoms that continue beyond 3 months after being infected will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Allergic rhinitis symptom control | 180 days
  Patients are free from any symptoms or reduction in the severity of the symptoms of allergic rhinitis.
  Total Nasal Symptom Score (TNSS) tool will be used for patients to self-rate their nasal symptoms, including nasal obstruction, itching, sneezing, secretion, runny nose, and sleep difficulty, on a 4-point Likert scale ranging from 0 (no symptom) to 3 (severe symptom). The scores will be summed; a higher score indicates the more severe the symptoms are. The measurement of nasal symptoms will be conducted at baseline, on Day 60 ±7, Day 120 ±7, and Day 180 ±7.
  The outcomes will be generated as a mean and standard deviation. A two-way repeated measure ANOVA analysis will be employed to determine the mean difference between the scores of the control group and the interventional group to determine the overall effectiveness of the intervention.

SECONDARY OUTCOMES:
Medication adherence to the allergic rhinitis treatment | 180 days
  It involved assessments of the patient's adherence to the intranasal corticosteroid treatment for allergic rhinitis.
  Medication adherence is measured by using a self-developed diary card. Patients will be asked to record their medication adherence levels on their daily use of intranasal corticosteroids.
  The measurement of adherence will be conducted on Day 60 ±7, Day 120 ±7, and Day 180 ±7.
  The estimation of the number of days that the patients declare that they are taking the medication will be summed for each measurement. A mean number of days of intranasal corticosteroid usage will be generated.
  A two-way repeated measure ANOVA analysis will be used to compare the between-group differences for the mean number of days of intranasal corticosteroid usage. A one-way repeated measure ANOVA analysis will be performed to determine within the group analysis. A value of P < 0.05 is considered statistically significant.
Improvement in quality of life of the allergic rhinitis patients | 180 days
  The 5-level EQ-5D version (EQ-5D-5L) questionnaire to assess the quality of life. It comprises a descriptive system and the EQ VAS (Visual Analogue Scale).
  The descriptive system comprises 5 dimensions, each with 5 response levels: no difficulties, slight, moderate, severe, and extreme problems. The outcome will be presented in a mean score and standard deviation in EQ-5D-5L utility index scores using the EQ-5D-5L index calculator for Malaysia.
  The EQ VAS captures the patients' total present health on a vertical visual analogue scale labelled "The best health you can imagine" (Max score: 100) and "The worst health you can imagine." (Min score: 0). EQ-5D VAS will be generated in a mean score and standard deviation.
  EQ-5D-5L will be measured at baseline, on Day 60 ±7, Day 120 ±7, and Day 180 ±7.
  A two-way repeated measure ANOVA analysis will be employed to determine the mean difference between the scores of the control and interventional groups.
Patients' knowledge of allergic rhinitis | 180 days
  Assessment of the patient's understanding of the symptoms and treatment of allergic rhinitis
  A self-administered questionnaire evaluating the knowledge on patients' understanding of intranasal corticosteroids. It consists of four items, and patients are required to answer each item by marking the responses as "yes", "no", or "unsure".
  The "yes" answer will be given a score of two; the "no" answer will be given a zero score, and the "not sure" will be given a score of one.
  The patients' knowledge will be assessed during the baseline data collection and on Day 180 ±7.
  The outcome will be presented in the mean score and standard deviation. Each question will be analysed separately. Between-group comparisons will be analysed using a T-test to compare the mean score difference between the two groups. Meanwhile, within-group comparisons will be analysed using the Paired T-test. A value of P < 0.05 is considered statistically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Raja Permaisuri Bainun Hospital, Ipoh, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chew CC, Chang CT, Lim XJ, Yong WY, George D, Letchumanan P, Rajan P, Chong CP. The management of allergic rhinitis by pharmacists in public services: a proposed PhaRmacISt-led Education Model (AR-PRISE). J Pharm Policy Pract. 2022 Nov 8;15(1):80. doi: 10.1186/s40545-022-00477-1. PMID 36348443
- [Result] Cvetkovski B, Kritikos V, Tan R, Yan K, Azzi E, Srour P, Bosnic-Anticevich S. A qualitative investigation of the allergic rhinitis network from the perspective of the patient. NPJ Prim Care Respir Med. 2019 Sep 19;29(1):35. doi: 10.1038/s41533-019-0147-5. PMID 31537804
- [Result] Members of the Workshops. ARIA in the pharmacy: management of allergic rhinitis symptoms in the pharmacy. Allergic rhinitis and its impact on asthma. Allergy. 2004 Apr;59(4):373-87. doi: 10.1111/j.1398-9995.2003.00468.x. No abstract available. PMID 15005760
- [Result] Bosnic-Anticevich S, Costa E, Menditto E, Lourenco O, Novellino E, Bialek S, Briedis V, Buonaiuto R, Chrystyn H, Cvetkovski B, Di Capua S, Kritikos V, Mair A, Orlando V, Paulino E, Salimaki J, Soderlund R, Tan R, Williams DM, Wroczynski P, Agache I, Ansotegui IJ, Anto JM, Bedbrook A, Bachert C, Bewick M, Bindslev-Jensen C, Brozek JL, Canonica GW, Cardona V, Carr W, Casale TB, Chavannes NH, Correia de Sousa J, Cruz AA, Czarlewski W, De Carlo G, Demoly P, Devillier P, Dykewicz MS, Gaga M, El-Gamal Y, Fonseca J, Fokkens WJ, Guzman MA, Haahtela T, Hellings PW, Illario M, Ivancevich JC, Just J, Kaidashev I, Khaitov M, Khaltaev N, Keil T, Klimek L, Kowalski ML, Kuna P, Kvedariene V, Larenas-Linnemann DE, Laune D, Le LTT, Lodrup Carlsen KC, Mahboub B, Maier D, Malva J, Manning PJ, Morais-Almeida M, Mosges R, Mullol J, Munter L, Murray R, Naclerio R, Namazova-Baranova L, Nekam K, Nyembue TD, Okubo K, O'Hehir RE, Ohta K, Okamoto Y, Onorato GL, Palkonen S, Panzner P, Papadopoulos NG, Park HS, Pawankar R, Pfaar O, Phillips J, Plavec D, Popov TA, Potter PC, Prokopakis EP, Roller-Wirnsberger RE, Rottem M, Ryan D, Samolinski B, Sanchez-Borges M, Schunemann HJ, Sheikh A, Sisul JC, Somekh D, Stellato C, To T, Todo-Bom AM, Tomazic PV, Toppila-Salmi S, Valero A, Valiulis A, Valovirta E, Ventura MT, Wagenmann M, Wallace D, Waserman S, Wickman M, Yiallouros PK, Yorgancioglu A, Yusuf OM, Zar HJ, Zernotti ME, Zhang L, Zidarn M, Zuberbier T, Bousquet J. ARIA pharmacy 2018 "Allergic rhinitis care pathways for community pharmacy": AIRWAYS ICPs initiative (European Innovation Partnership on Active and Healthy Ageing, DG CONNECT and DG Sante) POLLAR (Impact of Air POLLution on Asthma and Rhinitis) GARD Demonstration project. Allergy. 2019 Jul;74(7):1219-1236. doi: 10.1111/all.13701. Epub 2019 Apr 30. PMID 30565275
- [Result] Bousquet JJ, Schunemann HJ, Togias A, Erhola M, Hellings PW, Zuberbier T, Agache I, Ansotegui IJ, Anto JM, Bachert C, Becker S, Bedolla-Barajas M, Bewick M, Bosnic-Anticevich S, Bosse I, Boulet LP, Bourrez JM, Brusselle G, Chavannes N, Costa E, Cruz AA, Czarlewski W, Fokkens WJ, Fonseca JA, Gaga M, Haahtela T, Illario M, Klimek L, Kuna P, Kvedariene V, Le LTT, Larenas-Linnemann D, Laune D, Lourenco OM, Menditto E, Mullol J, Okamoto Y, Papadopoulos N, Pham-Thi N, Picard R, Pinnock H, Roche N, Roller-Wirnsberger RE, Rolland C, Samolinski B, Sheikh A, Toppila-Salmi S, Tsiligianni I, Valiulis A, Valovirta E, Vasankari T, Ventura MT, Walker S, Williams S, Akdis CA, Annesi-Maesano I, Arnavielhe S, Basagana X, Bateman E, Bedbrook A, Bennoor KS, Benveniste S, Bergmann KC, Bialek S, Billo N, Bindslev-Jensen C, Bjermer L, Blain H, Bonini M, Bonniaud P, Bouchard J, Briedis V, Brightling CE, Brozek J, Buhl R, Buonaiuto R, Canonica GW, Cardona V, Carriazo AM, Carr W, Cartier C, Casale T, Cecchi L, Cepeda Sarabia AM, Chkhartishvili E, Chu DK, Cingi C, Colgan E, de Sousa JC, Courbis AL, Custovic A, Cvetkosvki B, D'Amato G, da Silva J, Dantas C, Dokic D, Dauvilliers Y, Dedeu A, De Feo G, Devillier P, Di Capua S, Dykewickz M, Dubakiene R, Ebisawa M, El-Gamal Y, Eller E, Emuzyte R, Farrell J, Fink-Wagner A, Fiocchi A, Fontaine JF, Gemicioglu B, Schmid-Grendelmeir P, Gamkrelidze A, Garcia-Aymerich J, Gomez M, Gonzalez Diaz S, Gotua M, Guldemond NA, Guzman MA, Hajjam J, O'B Hourihane J, Humbert M, Iaccarino G, Ierodiakonou D, Illario M, Ivancevich JC, Joos G, Jung KS, Jutel M, Kaidashev I, Kalayci O, Kardas P, Keil T, Khaitov M, Khaltaev N, Kleine-Tebbe J, Kowalski ML, Kritikos V, Kull I, Leonardini L, Lieberman P, Lipworth B, Lodrup Carlsen KC, Loureiro CC, Louis R, Mair A, Marien G, Mahboub B, Malva J, Manning P, De Manuel Keenoy E, Marshall GD, Masjedi MR, Maspero JF, Mathieu-Dupas E, Matricardi PM, Melen E, Melo-Gomes E, Meltzer EO, Menditto E, Mercier J, Miculinic N, Mihaltan F, Milenkovic B, Moda G, Mogica-Martinez MD, Mohammad Y, Montefort S, Monti R, Morais-Almeida M, Mosges R, Munter L, Muraro A, Murray R, Naclerio R, Napoli L, Namazova-Baranova L, Neffen H, Nekam K, Neou A, Novellino E, Nyembue D, O'Hehir R, Ohta K, Okubo K, Onorato G, Ouedraogo S, Pali-Scholl I, Palkonen S, Panzner P, Park HS, Pepin JL, Pereira AM, Pfaar O, Paulino E, Phillips J, Picard R, Plavec D, Popov TA, Portejoie F, Price D, Prokopakis EP, Pugin B, Raciborski F, Rajabian-Soderlund R, Reitsma S, Rodo X, Romano A, Rosario N, Rottem M, Ryan D, Salimaki J, Sanchez-Borges MM, Sisul JC, Sole D, Somekh D, Sooronbaev T, Sova M, Spranger O, Stellato C, Stelmach R, Suppli Ulrik C, Thibaudon M, To T, Todo-Bom A, Tomazic PV, Valero AA, Valenta R, Valentin-Rostan M, van der Kleij R, Vandenplas O, Vezzani G, Viart F, Viegi G, Wallace D, Wagenmann M, Wang Y, Waserman S, Wickman M, Williams DM, Wong G, Wroczynski P, Yiallouros PK, Yorgancioglu A, Yusuf OM, Zar HJ, Zeng S, Zernotti M, Zhang L, Zhong NS, Zidarn M; ARIA Study Group; MASK Study Group. Next-generation ARIA care pathways for rhinitis and asthma: a model for multimorbid chronic diseases. Clin Transl Allergy. 2019 Sep 9;9:44. doi: 10.1186/s13601-019-0279-2. eCollection 2019. PMID 31516692
- [Result] Lourenco O, Bosnic-Anticevich S, Costa E, Fonseca JA, Menditto E, Cvetkovski B, Kritikos V, Tan R, Bedbrook A, Scheire S, Bachert C, Bialek S, Briedis V, Boussery K, Canonica GW, Haahtela T, Kuna P, Novellino E, Samolinski B, Schunemann HJ, Wallace D, Bousquet J. Managing Allergic Rhinitis in the Pharmacy: An ARIA Guide for Implementation in Practice. Pharmacy (Basel). 2020 May 16;8(2):85. doi: 10.3390/pharmacy8020085. PMID 32429362
- [Result] Jose J, Cvetkovski B, Kritikos V, Tan R, Bosnic-Anticevich S, Lourenco O. Interventions Delivered in the Community Pharmacy to Manage Allergic Rhinitis- A Systematic Review of the Literature. Pharmacy (Basel). 2020 May 6;8(2):80. doi: 10.3390/pharmacy8020080. PMID 32384674
- [Result] Arsoy G, Varis A, Saloumi LM, Abdi A, Basgut B. Insights on Allergic Rhinitis Management from a Northern Cyprus Perspective and Evaluation of the Impact of Pharmacist-Led Educational Intervention on Patients' Outcomes. Medicina (Kaunas). 2018 Nov 7;54(5):83. doi: 10.3390/medicina54050083. PMID 30405059
- [Result] Bousquet J, Schunemann HJ, Togias A, Bachert C, Erhola M, Hellings PW, Klimek L, Pfaar O, Wallace D, Ansotegui I, Agache I, Bedbrook A, Bergmann KC, Bewick M, Bonniaud P, Bosnic-Anticevich S, Bosse I, Bouchard J, Boulet LP, Brozek J, Brusselle G, Calderon MA, Canonica WG, Caraballo L, Cardona V, Casale T, Cecchi L, Chu DK, Costa EM, Cruz AA, Czarlewski W, D'Amato G, Devillier P, Dykewicz M, Ebisawa M, Fauquert JL, Fokkens WJ, Fonseca JA, Fontaine JF, Gemicioglu B, van Wijk RG, Haahtela T, Halken S, Ierodiakonou D, Iinuma T, Ivancevich JC, Jutel M, Kaidashev I, Khaitov M, Kalayci O, Kleine Tebbe J, Kowalski ML, Kuna P, Kvedariene V, La Grutta S, Larenas-Linnemann D, Lau S, Laune D, Le L, Lieberman P, Lodrup Carlsen KC, Lourenco O, Marien G, Carreiro-Martins P, Melen E, Menditto E, Neffen H, Mercier G, Mosgues R, Mullol J, Muraro A, Namazova L, Novellino E, O'Hehir R, Okamoto Y, Ohta K, Park HS, Panzner P, Passalacqua G, Pham-Thi N, Price D, Roberts G, Roche N, Rolland C, Rosario N, Ryan D, Samolinski B, Sanchez-Borges M, Scadding GK, Shamji MH, Sheikh A, Bom AT, Toppila-Salmi S, Tsiligianni I, Valentin-Rostan M, Valiulis A, Valovirta E, Ventura MT, Walker S, Waserman S, Yorgancioglu A, Zuberbier T; Allergic Rhinitis and Its Impact on Asthma Working Group. Next-generation Allergic Rhinitis and Its Impact on Asthma (ARIA) guidelines for allergic rhinitis based on Grading of Recommendations Assessment, Development and Evaluation (GRADE) and real-world evidence. J Allergy Clin Immunol. 2020 Jan;145(1):70-80.e3. doi: 10.1016/j.jaci.2019.06.049. Epub 2019 Oct 15. PMID 31627910
- [Result] Cvetkovski B, Tan R, Kritikos V, Yan K, Azzi E, Srour P, Bosnic-Anticevich S. A patient-centric analysis to identify key influences in allergic rhinitis management. NPJ Prim Care Respir Med. 2018 Sep 13;28(1):34. doi: 10.1038/s41533-018-0100-z. PMID 30213945
- [Derived] Chew CC, Lim XJ, Letchumanan P, Rajan P, Chong CP. Pharmacist-Led Education Intervention for Adults With Allergic Rhinitis: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2517160. doi: 10.1001/jamanetworkopen.2025.17160. PMID 40668584
- [Derived] Chew CC, Lim XJ, Letchumanan P, George D, Rajan P, Chong CP. The effectiveness of pharmacist-led educational model in adult patients with allergic rhinitis: a single-center randomized control trial protocol (AR-PRISE RCT). Trials. 2024 Apr 25;25(1):279. doi: 10.1186/s13063-024-08111-y. PMID 38664701